CLINICAL TRIAL: NCT02788214
Title: Helicobacter Pylori Genome Project (HpGP)
Status: Terminated | Type: Observational
Why Stopped: research determined not to be human subject research
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: New England Biolabs, USA (Unknown); National Institute of Infectious Diseases, Japan (Unknown); National Institute of Genetics, Japan (Unknown); Chiba University, Japan (Unknown); National Institute for Basic Biology, Japan (Unknown); Instituto Mexicano del Seguro Social (Other Government); Universidade de Lisboa, Portugal (Unknown); Instituto de Biomedicina de Valencia, Spain (Unknown); University of Bath, UK (Unknown); Vanderbilt University Medical Center, USA (Unknown); Karolinska Institutet (Other); University of Tokyo, Japan (Unknown); Max von Pettenkofer-Institute of Hygiene and Medical Microbiology, Germany (Unknown); Universidad de Chile, Chile (Unknown); HOSEI University, Japan (Unknown)
Responsible Party: Sponsor
Other Study IDs: NCI-2020-07069; 16-C-N120; 999916120 (Other: National Cancer Institute)
Record Dates: First submitted 2016-05-28; First posted 2016-06-02 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer; Non-Atrophic Gastritis; Intestinal Metaplasia
Keywords: Gastric Cancer; Bacterial Risk Factors; DNA Methylation; DNA Sequencing; Biobank; Helicobacter pylori; SMRT/PacBio
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Helicobacter pylori strains.

GROUPS / COHORTS (3):
- Advanced intestinal metaplasia: H. pylori strains from patients with:
  * Complete-type intestinal metaplasia with extension to corpus, or
  * Incomplete-type intestinal metaplasia of any extent
- Non-atrophic gastritis: H. pylori strains from patients with non-atrophic gastritis
- Gastric cancer: H. pylori strains from patients with gastric cancer

SUMMARY:
Helicobacter pylori is a common bacterial infection. It can lead to severe stomach problems, including stomach cancer. Researchers want to look at samples of the bacteria. These H. pylori strains will be taken from chronically infected people. They want to identify the genetic and epigenetic differences in H. pylori strains. This could help predict which people who get infected with the bacteria will get stomach cancer. This could lead to the cancer being detected earlier. It could also mean less people get stomach cancer.

Objectives:

To study genetic variations of H. pylori strains based on samples from chronically infected people. To identify the features of strains that might lead to severe stomach problems or stomach cancer.

Eligibility:

People ages 30-70 years who need an upper endoscopy or who were recently diagnosed with stomach cancer

Design:

Participants will be screened by the doctor who does their procedure and a study nurse.

Participants who have endoscopy will have ~6 biopsies removed. These are tissue samples. They are about the size of a grain of rice. Participants will allow the study team to access reports from their stomach exam.

Participants with stomach cancer will donate some of the tissue that will be removed during their clinical care. They will allow the study team to access reports of their surgery. They will also allow them to access the microscope slides of their stomach.

DETAILED DESCRIPTION:
Helicobacter pylori, a Gram-negative bacterium associated with a spectrum of benign and malignant gastric conditions, is one of the most genetically variable pathogens. Variations in a few genes have been associated with risk of inflammation and carcinogenesis, but to date no systematic study has evaluated the entire bacterial genome. We propose a multicountry study to establish and analyze an informative international collection of H. pylori clinical isolates from residents of defined geographic areas. Molecular characterization will be conducted at the NCI/DCEG. Our hypothesis is that genetic and epigenetic variations in H. pylori strains among chronically infected individuals may affect risk of progression to gastric cancer. Findings from this study may help to characterize the differential virulence among H. pylori isolates and suggest predictive biomarkers for early diagnosis of cancer. The bacterial isolates and databases from this study will also provide a foundation for further elucidation of H. pylori pathogenesis.

ELIGIBILITY:
INCLUSION CRITERIA:

H. pylori strains collected from:

1. Adult aged 30 to 70 years old.
2. Patients who need upper endoscopy (examination of the lining of their stomach with a flexible tube).
3. Patients with stomach cancer.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori strains from patients with various gastrointestinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Bacterial DNA sequence | At enrollment
  genome and methylome

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Rabkin, M.D., Principal Investigator — National Cancer Institute (NCI); M. Constanza Camargo, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (94):
- United States (7):
  - White River Medical Center, Batesville, Arkansas
  - Stanford University, Stanford, California
  - Georgia Cancer Center Biorepository, Athens, Georgia
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Albert Einstein College of Medicine, The Bronx, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Université Ferhat Abbas, Sétif, Algeria
- Hospital Alemán, Buenos Aires, Argentina
- Dhaka Medical College and Hospital, Dhaka, Bangladesh
- Ghent University, Ghent, Belgium
- Brazil (2):
  - Universidade Federal de Minas Gerais, Belo Horizonte
  - AC Camargo Cancer Center, São Paulo
- Bulgaria (2):
  - Medical University of Sofia, Sofia
  - Tsaritsa Yoanna University Hospital, Sofia
- Defence Services General Hospital, Yangon, Burma
- University of Dschang, Dschang, Cameroon
- University of Alberta, Edmonton, Canada
- Chile (3):
  - Universidad de Concepción, Concepción
  - Hospital Hanga Roa, Easter Island
  - Pontificia Universidad Catolica, Santiago
- Colombia (3):
  - Instituto Nacional de Cancerología, Bogotá
  - Universidad del Valle, Cali
  - Universidad de Nariño, Pasto
- Universidad de Costa Rica, San José, Costa Rica
- Democratic Republic of the Congo (2):
  - University of Kinshasa, Kinshasa
  - University of Mbuji Mayi, Mbuji-Mayi
- Universidad Autónoma de Santo Domingo, Santo Domingo, Dominican Republic
- C.H.U. Pellegrin, Bordeaux, France
- Otto-von-Guericke Universitätsklinikum, Magdeburg, Germany
- University of Cape Coast, Cape Coast, Ghana
- Greece (2):
  - Evangelismos Hospital and Hellenic Pasteur Institute, Athens
  - Hellenic Pasteur Institute, Athens
- Universidad San Carlos, Guatemala City, Guatemala
- Hospital de Occidente, Santa Rosa de Copán, Honduras
- National University Hospital, Reykjavik, Iceland
- Kasturba Medical College Manipal, Manipal, India
- Indonesia (2):
  - University of Indonesia, Depok
  - Universitas Airlangga, Surabaya
- Digestive Disease Research Institute, Tehran, Iran
- Bar Ilan University, Ramat Gan, Israel
- Centro di Rferimento Oncologico, Aviano, Italy
- Japan (5):
  - Nagoya City University, Nagoya
  - Oita University, Ōita
  - HOSEI University, Tokyo
  - Kyorin University, Tokyo
  - Nippon Medical School, Tokyo
- Jordan University of Science and Technology, Ar Ramtha, Jordan
- Central Asian Cancer Institute, Almaty, Kazakhstan
- Tenwek Hospital, Bomet, Kenya
- Kyrgyz State Medical Academy, Bishkek, Kyrgyzstan
- University of Latvia, Riga, Latvia
- Lithuanian University of Health Sciences, Kaunas, Lithuania
- University of Malaya, Kuala Lumpur, Malaysia
- Instituto Nacional de Cancerología, Mexico City, Mexico
- Nepal (2):
  - Chitwan Medical College, Bharatpur
  - Tribhuvan University Teaching Hospital, Kathmandu
- Nigeria (5):
  - University of Calabar Teaching Hospital, Calabar
  - University of Nigeria Teaching Hospital, Enugu
  - Babcock Universtiy Teaching Hospital, Ilishan
  - University of Jos / University Teaching Hospital, Jos
  - Federal Medical Center, Lagos
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Universidad Peruana Cayetano Heredia, Lima
- Poland (2):
  - University of Lublin, Publin
  - Wroclaw Medical Center, Wroclaw
- Portugal (2):
  - Instituto Nacional de Saúde Dr. Ricardo Jorge, Lisbon
  - University of Porto, Porto
- University of Puerto Rico, San Juan, Puerto Rico
- Clinical Research Center of Moscow, Moscow, Russia
- National University Hospital, Singapore, Singapore
- Chris Hani Baragwanath Academic Hospital, Soweto, South Africa
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Chung-Ang University Hospital, Seoul
  - National Cancer Center, Seoul
- Spain (12):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General de Granollers, Barcelona
  - Hospital Universitari Parc Tauli, Barcelona
  - Institut d'Investigació Biomédica de Bellvitge (Idibell), Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital de Leon, León
  - Hospital de la Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Lozano Blesa University Hospital, Zaragoza
- Sudan University of Science and Technology, Khartoum, Sudan
- Karolinska Institutet, Stockholm, Sweden
- Switzerland (2):
  - University of Bern, Bern
  - University of Zurich, Zurich
- National Taiwan University Hospital, Taipei, Taiwan
- Istanbul University, Istanbul, Turkey (Türkiye)
- Cho Ray Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Correa P, Haenszel W, Cuello C, Tannenbaum S, Archer M. A model for gastric cancer epidemiology. Lancet. 1975 Jul 12;2(7924):58-60. doi: 10.1016/s0140-6736(75)90498-5. PMID 49653
- [Background] Tomb JF, White O, Kerlavage AR, Clayton RA, Sutton GG, Fleischmann RD, Ketchum KA, Klenk HP, Gill S, Dougherty BA, Nelson K, Quackenbush J, Zhou L, Kirkness EF, Peterson S, Loftus B, Richardson D, Dodson R, Khalak HG, Glodek A, McKenney K, Fitzegerald LM, Lee N, Adams MD, Hickey EK, Berg DE, Gocayne JD, Utterback TR, Peterson JD, Kelley JM, Cotton MD, Weidman JM, Fujii C, Bowman C, Watthey L, Wallin E, Hayes WS, Borodovsky M, Karp PD, Smith HO, Fraser CM, Venter JC. The complete genome sequence of the gastric pathogen Helicobacter pylori. Nature. 1997 Aug 7;388(6642):539-47. doi: 10.1038/41483. PMID 9252185
- [Background] Krebes J, Morgan RD, Bunk B, Sproer C, Luong K, Parusel R, Anton BP, Konig C, Josenhans C, Overmann J, Roberts RJ, Korlach J, Suerbaum S. The complex methylome of the human gastric pathogen Helicobacter pylori. Nucleic Acids Res. 2014 Feb;42(4):2415-32. doi: 10.1093/nar/gkt1201. Epub 2013 Dec 2. PMID 24302578
- See also: HpGP webpage — https://dceg.cancer.gov/research/how-we-study/genomic-studies/h-pylori-genome-project